CLINICAL TRIAL: NCT05470920
Title: Randomized, Controlled Trial of an Electronic Decision Aid for Genetic Testing in Inherited Cancer Syndromes
Brief Title: Genetic Testing Decision Aid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Daniel C Chung, Principal Investigator, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 22-155; U01CA243695 (NIH)
Record Dates: First submitted 2022-07-15; First posted 2022-07-22 (Actual); Last update posted 2025-08-13 (Actual); Status verified 2025-08

CONDITIONS: Epithelial Ovarian Carcinoma; Pancreas Adenocarcinoma
Keywords: pancreas adenocarcinoma.; epithelial ovarian carcinoma; decision aid; inherited cancer syndrome; genetic testing
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial; Neoplastic Syndromes, Hereditary

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Electronic decision aid arm (Experimental): Receive decision aid followed by an appointment with their oncologist.
  Interventions: Behavioral: Electronic Decision Aid
- Genetic counselor Arm (Active Comparator): Receive pretest counseling with a genetic counselor.
  Interventions: Behavioral: Pre-Test Genetic Counseling

INTERVENTIONS:
Behavioral: Electronic Decision Aid — Decision aid followed by an appointment with an oncologist. Will complete surveys/questionnaires
  Arms: Electronic decision aid arm
Behavioral: Pre-Test Genetic Counseling — Receive pretest counseling with a genetic counselor. Will complete surveys/questionnaires
  Arms: Genetic counselor Arm

SUMMARY:
This is a randomized trial to evaluate the effectiveness of an electronic decision aid tool versus a traditional genetic counselor session for multi-gene panel testing for people with ovarian or pancreatic cancer

DETAILED DESCRIPTION:
The research study procedures include: screening for eligibility and study questionnaires that would be performed in conjunction with either the genetic counselor visit or use of the electronic decision aid. The study questionnaires include:

* Knowledge Survey
* Shared Decision Making Process Survey
* Decisional Conflict Scale

The research study will last up to 2 weeks. It is expected that about 350 people will take part in this research study.

The National Cancer Institute (NCI) is supporting this research study by providing funding for the research

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* Being seen in clinic at Massachusetts General Hospital or Boston Medical Center
* Diagnosed with malignant epithelial ovarian carcinoma or malignant pancreatic adenocarcinoma.

Exclusion Criteria :

* Unable or unwilling to provide informed consent, undergo randomization, or complete the surveys associated with the study
* Previous germline genetic testing
* History of hereditary pancreatitis
* Members of the following vulnerable populations: adults unable to consent, individuals who are not yet adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2022-10-14 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Average change in knowledge survey score | baseline (prior to participant completing either genetics sessions) to 1-week following session, approximately 2 weeks
  Average change in score on a 10-question knowledge survey to assess basic information about genetics and genetic testing that was covered in their appointment. Scores on the scale range from 0-10. Higher values in the change in knowledge survey score suggest greater amount of knowledge gained in the genetics session.
Decisional Conflict Scores | 1 week after genetics session
  The decisional conflict score is a score ranging from 0-100 that is measured from a 10-question validated decisional conflict scale. The scale assesses participant's confidence in their decision with higher scores indicating higher decisional conflict.
Shared Decision Making Process Scores | 1 week after genetics session
  The shared decision making process score is a score on a scale of 1-4 based on responses on a validated 4-item shared-decision making scale. The scale assesses how well the decision aid/oncology provider, or the genetic counselor engaged in shared decision-making as perceived by the subject. Higher scores on this scale indicate more shared decision making.

SECONDARY OUTCOMES:
Average time between genetic testing recommendation and sample collection | Initial recorded recommendation/referral for genetic testing until the date of sample collection, assessed up to 6 months
  Difference between the two study arms in the time it takes between participants being recommended for genetic testing and a sample being collected.
Average Duration of Decision Making Process | Approximately 30 minutes - 1 hour
  Amount of time patients spend learning and making a decision about genetic testing in both arms of the study.
Ratio of the number of participants who chose each of the three panels offered | At the conclusion of genetics session (day 1)
  Ratios of participants who choose the small, intermediate, and broad testing panel in both arms of the study.
Percentage of participants choosing genetic testing | At the conclusion of genetics session (day 1)
  Percentage of participants in each arm of the study who choose to get genetic testing after the educational intervention

CONTACTS AND LOCATIONS:
Overall Officials: Daniel C. Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mass General at North Shore Cancer Center, Danvers, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation